CLINICAL TRIAL: NCT05256797
Title: Prediction of the COBRRA AF Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-COBRRA-AF
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rivaroxaban: Reference group
  Interventions: Drug: Rivaroxaban
- Apixaban: Exposure group
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Rivaroxaban — Any rivaroxaban dispensing claim is used as the reference group
  Other Names: Xarelto
  Groups: Rivaroxaban
Drug: Apixaban — Any apixaban dispensing claim is used as the exposure group
  Other Names: Eliquis
  Groups: Apixaban

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Non-valvular atrial fibrillation

Exclusion Criteria:

* Prior anticoagulant use [Day -180, Day 0]
* Stage 4 or 5 chronic kidney disease or end-stage renal disease [Day -180, Day 0]
* Dialysis or renal transplant [Day -180, Day 0]
* Recent major or clinically relevant non-major bleeding [Day -180, Day 0]
* Other indications for anticoagulation (DVT, PE, or prosthetic heart valve) [Day -180, Day 0]
* Use of an antiplatelet [Day -180, Day 0]
* Significant liver disease and coagulopathy [Day -180, Day 0]
* Use of CYP3A4 or P-gp inhibitors or inducers [Day -180, Day 0]
* Pregnancy or breastfeeding [Day -180, Day 0]
* Cancer [Day -180, Day 0]
* Bypass surgery, obesity, or the use of a weight loss or appetite suppressor [Day -180, Day 0]
* Mitral stenosis with or without insufficiency, mitral rheumatic insufficiency, and other/unspecified mitral valve disorders [Day -180, Day 0]

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban to apixaban users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of rivaroxaban or apixaban (index date). Analysis is restricted to patients with non-valvular atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 353980 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivaroxaban | Apixaban
Started | 176990 | 176990
Completed | 176990 | 176990
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Apixaban | Total
Number analyzed (Participants) | 176,990 | 176,990 | 353980
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26,276 | 26,331 | 52607
  >=65 years | 150,714 | 150,659 | 301373
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.91 (9.65) | 73.88 (9.75) | 73.90 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88,058 | 88,018 | 176076
  Male | 88,932 | 88,972 | 177904
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 127,937 | 127,949 | 255886
  Asian | 2,554 | 2,554 | 5108
  Black | 7,016 | 7,011 | 14027
  Hispanic | 4,140 | 4,162 | 8302
  North American Native | 326 | 332 | 658
  Other | 1,283 | 1,283 | 2566
  Unknown/Missing | 2,830 | 2,792 | 5622
  N/A | 30,904 | 30,907 | 61811
Region of Enrollment [Number; unit: participants]
  United States | 176,990 | 176,990 | 353980

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Major Bleeding or Clinically Relevant Non-major Bleeding Events
Description: Claims-based algorithm: incidence of major bleeding or clinically relevant non-major bleeding events
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 9.2 [9.0 to 9.5] | 6.4 [6.2 to 6.6]
Statistical Analysis 1: Comparison: Rivaroxaban vs Apixaban; Hazard ratio; Test type: Superiority; Cox Proportional Hazard = 0.69, 95% CI 2-sided [0.66 to 0.71]

2. Secondary Outcome: Incidence of Major Bleeding
Description: Claims-based algorithm: Incidence of major bleeding
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 4.0 [3.8 to 4.1] | 2.4 [2.3 to 2.5]

3. Secondary Outcome: Incidence of Clinically Relevant Non-major Bleeding
Description: Claims-based algorithm: Incidence of clinically relevant non-major bleeding
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 8.7 [8.4 to 8.9] | 5.9 [5.8 to 6.1]

4. Secondary Outcome: Incidence of All-cause Mortality
Description: Claims-based algorithm: Incidence of all-cause mortality
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 2.7 [2.6 to 2.8] | 2.4 [2.3 to 2.5]

5. Secondary Outcome: Incidence of Stroke
Description: Claims-based algorithm: Incidence of stroke
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 1.1 [1.0 to 1.2] | 0.9 [0.8 to 1.0]

6. Secondary Outcome: Incidence of Extracranial Bleeding
Description: Claims-based algorithm: Incidence of extracranial bleeding (any position)
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 3.6 [3.5 to 3.8] | 2.1 [2.0 to 2.2]

7. Secondary Outcome: Incidence of Intracranial Bleeding
Description: Claims-based algorithm: Incidence of intracranial bleeding (any position)
Time Frame: Through study completion or censoring, up to 365 days
Population: Propensity score matched. population across 3 databases
Measure: Number (95% Confidence Interval); unit: No. of new events per 100 person-years
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 176990 | 176990
No. of new events per 100 person-years | 0.4 [0.3 to 0.4] | 0.3 [0.3 to 0.4]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed from enrollment to completion of study, up to 365 days
Description: Only All-Cause Mortality was monitored/assessed. Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Rivaroxaban | Apixaban
All-Cause Mortality (participants affected / at risk) | 1958/176990 | 1840/176990
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05256797/Prot_002.pdf